CLINICAL TRIAL: NCT00565656
Title: A Phase II Trial of Bevacizumab in Myelodysplastic Syndromes (Int-1, Int-2 and High Risk According to IPSS) With Excess of Marrow Blasts
Brief Title: A Trial of Bevacizumab in Myelodysplastic Syndromes (Int-1, Int-2 and High Risk According to International Prognostic Scoring System (IPSS)) With Excess of Marrow Blasts
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-PP-05; AFSSAPS number:060748
Record Dates: First submitted 2007-11-28; First posted 2007-11-30 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2009-06

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic syndromes (int-1, int-2 and high risk according to IPSS) with excess of marrow blasts including CMML with leucocytes<10 000/mm3
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Bevacizumab
  Interventions: Drug: BEVACIZUMAB

INTERVENTIONS:
Drug: BEVACIZUMAB — Administration of Bevacizumab

SUMMARY:
The objectives of this phase II trial are to test the efficacy and tolerance of Bevacizumab in MDS patients with excess of marrow blasts and to evaluate the impact of Bevacizumab on angiogenesis and erythropoiesis.

To limit the myelotoxicity observed in the preliminary phase II study, Bevacizumab will be administrated at the initial dose of 5 mg/kg.

The primary endpoint will be response: Complete Remission (CR), Partial Remission (PR) and hematological improvement (HI) according to IWG criteria (see appendix 3).

The secondary endpoints will be survival, response duration, side effects, evaluation of angiogenesis (bone marrow microvessel density, VEGF plasma level, VEGF mRNA expression, HIF-1alpha expression).

The design of this study consists of three study periods: pre-treatment (screening), treatment (loading and maintenance), and follow-up. All patients will participate in the study for at least 12 weeks of therapy, a 4-week follow-up visit, and long-term follow-up unless the criteria for planned or unplanned early discontinuation are met.

ELIGIBILITY:
Inclusion Criteria:

* MDS patient with excess of marrow blasts (≥ 5%) including RAEB, RAEB-t and CMML with leucocytes < 10 000/mm3 according to FAB classification
* IPSS int-1, int-2 or high
* Age > 60 years (younger adults may be included, but only in the absence of donor for allogeneic stem cell transplantation, and if contra-indication to intensive chemotherapy)
* No previous allogeneic SCT or intensive anthracycline-Ara C chemotherapy.
* Adequate renal function:

  * Serum creatinine ≤ 1.25 x ULN or calculated creatinine clearance ≥ 50 mL/min AND
  * Urine dipstick for proteinuria < 2+. Patients discovered to have ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1 g of protein in 24 hours
* Adequate liver function:

  * Total bilirubin < 1.5 x upper limit of normal (ULN) AND Asparagine aminotransferase (AST), alanine aminotransferase (ALT) < 2.5 x ULN in patients without liver metastases
* International normalised ratio (INR) ≤1.5 and prothrombin time (PPT) ≤ 1.5 x ULN within 7 days prior to enrolment
* If female, should not be pregnant or breast-feeding. Women with an intact uterus (unless amenorrhoeic for the last 24 months) must have a negative serum pregnancy test within 28 days prior to enrollment into the study. If a serum pregnancy test is not performed within 7 days prior to the first dose of bevacizumab, a confirmatory urine test (within 7 days prior to the first dose of bevacizumab) is required.
* Life expectancy ≥ 6 months
* Patient with health insurance
* Written informed consent

Exclusion Criteria:

* Therapy related MDS (after chemo or radiotherapy) for a previous neoplasm or other disease including AML
* A preexisting thrombocytopenia < 20 000/mm3
* Major surgery (including open biopsy), significant traumatic injury within 28 days prior to enrolment or anticipation of the need for major surgery during study treatment
* Minor surgery, including insertion of an indwelling catheter, within 24 hours prior to the first bevacizumab infusion
* Prior tumor (except localized cervix carcinoma or cutaneous basal cell carcinoma) unless in remission for at least 3 years.
* Uncontrolled diabetes mellitus
* Current or recent (within 10 days of first dose of bevacizumab) use of aspirin (> 325 mg/day)
* Uncontrolled hypertension (blood pressures: systolic > 150 mmHg and/or diastolic > 100 mmHg)
* Clinically significant (i.e., active) cardiovascular disease for example CVA (≤6 months before enrollment), myocardial infarction (≤ 6 months before enrollment), unstable angina, congestive heart failure NYHA Class ≥ II, serious cardiac arrhythmia requiring medication during the study and might interfere with regularity of the study treatment, or not controlled by medication
* Non-healing wound, active peptic ulcer or bone fracture
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months of enrolment
* Women with an intact uterus (unless amenorrhoeic for the last 24 months) not using effective, non-hormonal means of contraception (intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly or surgically sterile) during the study and for a period of 6 months following the last administration of bevacizumab. Men who do not agree to use effective contraception during the study and for a period of 60 days following the last administration of bevacizumab
* Investigational treatment for MDS within 6 weeks of treatment onset
* Patients unable to give informed consent or to be followed up adequately
* Known hypersensitivity to a product from Chinese Hamster Ovary mammalian cell or to a recombinant humanized monoclonal antibody

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Bone marrow evaluation Peripheral blood evaluation Cytogenetic response Hematologic improvement (HI) | Before the first injection, weekly during twenty weeks and four weeks after the last injection

SECONDARY OUTCOMES:
The secondary endpoints will be survival, side effects | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Laurence LEGROS, Doctor, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (10):
- France (10):
  - Department of clinical hematology, Avignon
  - Department of Hematology, Bobigny
  - Department of Hematology, Lyon
  - Paoli-Calmette Institut, Marseille
  - Department of Clinical hematology, Archet Hospital, CHU de Nice, Nice
  - Department of Onco-Hematology, Caremeau Hospital, CHU Nîmes, Nîmes
  - Department of clinical hematology, Robert Debré Hospital, Reims
  - Department of Hematology and Oncology, CHU de Strasbourg, Strasbourg
  - Service de Médecine Interne, Toulouse
  - Department of clinical hematology, Vandœuvre-lès-Nancy